CLINICAL TRIAL: NCT03278743
Title: Higher Tea Consumption is Associated With Better Performance on Measures of Attention and Psychomotor Speed in the Very Old: The Newcastle 85+ Study
Brief Title: Tea Consumption and Cognitive Performance in the Very Old
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: UNewcastle
Record Dates: First submitted 2017-08-14; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Cognition
Keywords: tea; cognition; very old; Newcastle 85+; epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low to moderate tea consumption: consumption of 0.4 to 4.6 cups of tea (200 ml) per day (n=463)
  Interventions: Other: Cognitive performance and cognitive decline
- High tea consumption: consumption of 4.6 to 11.9 cups of tea (200 ml) per day (n=213)
  Interventions: Other: Cognitive performance and cognitive decline

INTERVENTIONS:
Other: Cognitive performance and cognitive decline — Assess the global and domain specific (memory, speed and attention) cognitive function at baseline and over 5 years in the high vs. low/moderate tea consumption groups

SUMMARY:
Studies have found a beneficial effect of tea consumption on the reduction of risk of cognitive impairment and dementia in older aged populations. However, there is a paucity of data on these associations in the very old defined as individuals aged 85 years and over. Therefore, we hypothesized that higher tea consumption was associated with better global and domain-specific cognitive function. We investigated the relationship between tea consumption in the very old and measures of global cognitive function, memory, attention and psychomotor speed.

The Newcastle 85+ Study was a longitudinal (5-years), population-based cohort study of individuals aged 85+ years in North East England, United Kingdom. The final sample included 676 community-dwelling and institutionalized men and women recruited through general medical practices.

Baseline tea consumption was assessed through a 2x24-hr multiple pass recall and longitudinal measures of global and domain specific (memory, speed and attention) cognitive function through the standardized mini-mental state examination and the cognitive drug research system. Linear mixed models, controlling for demographic (e.g. age, sex and education) and health variables were used to determine whether tea consumption was protective against cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Born in 1921
* Permanently registered with a participating general practice in Newcastle upon Tyne or North Tyneside primary care trusts in the UK

Exclusion Criteria:

* End-stage illness
* Individuals who might pose a safety risk to a nurse visiting alone, with dementia
* Clinical diagnosis of dementia at baseline

Ages: 85 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling and institutionalized men and women recruited through general medical practices in North East England, UK (n=676) and born in 1921 (85 years old at baseline).
Sampling Method: Non-Probability Sample
Enrollment: 1042 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Standardized mini-mental state examination | Baseline
  Measure of global cognition (Score 0-30)
Rate of decline of the standardized mini-mental state examination | Baseline to 5 years follow-up
  Measure of global cognition (Score 0-30)

SECONDARY OUTCOMES:
Simple reaction time | Baseline
  Simple reaction time assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box. The participant is instructed to press "YES" as quickly as possible every time the word "YES" is presented on the screen. In total, 30 "YES" stimuli are presented with varying inter-stimulus interval. (ms)
Rate of reaction speed decline | Baseline to 3 years follow-up
  Simple reaction time assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box.The participant is instructed to press "YES" as quickly as possible every time the word "YES" is presented on the screen. In total, 30 "YES" stimuli are presented with varying inter-stimulus interval. (ms)
Choice reaction time | Baseline
  Choice reaction time assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box. Either the word "YES" or "NO" is presented on the screen and the participant is instructed to press the corresponding button as quickly as possible. There are 30 trials for each stimulus word, which is chosen randomly with equal probability, with varying inter-stimulus interval. (ms)
Rate of reaction choice decline | Baseline to 3 years follow-up
  Choice reaction time assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box.Either the word "YES" or "NO" is presented on the screen and the participant is instructed to press the corresponding button as quickly as possible. There are 30 trials for each stimulus word, which is chosen randomly with equal probability, with varying inter-stimulus interval. (ms)
Digit vigilance task | Baseline
  Digit vigilance task assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box. Target digit is randomly selected and constantly displayed to the right of the screen. A series of digits (0-9) are presented in the centre of the screen at the rate of 150 per minute. The participant is required to press the "YES" button as quickly as possible every time the digit in the series matches the target digit. There are 300 digits in the series and the task lasts for 2 minutes. (ms)
Rate of digit vigilance task decline | Baseline to 3 years follow-up
  Digit vigilance task assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box. Target digit is randomly selected and constantly displayed to the right of the screen. A series of digits (0-9) are presented in the centre of the screen at the rate of 150 per minute. The participant is required to press the "YES" button as quickly as possible every time the digit in the series matches the target digit. There are 300 digits in the series and the task lasts for 2 minutes. (ms)
Word recognition | Baseline
  Word recognition was assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box. A list of words is presented on screen for the subject to remember. Immediately after the presentation the subject is asked to recall as many words as possible. 20 minutes later, the same list of words is presented with added distracter words. For each word, the subject is asked to indicate whether or not it belongs o the original list by pressing 'YES' or 'NO'.
Rate of word recognition decline | Baseline to 3 years follow-up
  Word recognition was assessed using the Cognitive Drug Research (CDR) computerised system. The CDR tasks were presented on a hi-resolution Windows-based laptop computer (Motion Computing LE1600 Tablet PC with keyboard accessory) and participants responded using a two-button (NO/YES) response box.A list of words is presented on screen for the subject to remember. Immediately after the presentation the subject is asked to recall as many words as possible. 20 minutes later, the same list of words is presented with added distracter words. For each word, the subject is asked to indicate whether or not it belongs to the original list by pressing 'YES' or 'NO'.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Kirkwood, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Data request
URL: http://research.ncl.ac.uk/85plus/datarequests/